CLINICAL TRIAL: NCT00991016
Title: A Phase 1 Randomized, Double Blind (3rd Party Open), Placebo Controlled Combined Single And Multiple Dose Safety, Tolerability And Pharmacokinetics Study Of Orally Administered PF-04805712 In Healthy Volunteers
Brief Title: Single and Multiple Dose Safety, Tolerability, and Pharmacokinetics Study of PF-04805712 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: B1411001 was terminated after completion of 4 cohorts of the multiple ascending dose phase, as additional data were deemed unnecessary. No safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1411001
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04805712 (Experimental)
  Interventions: Drug: PF-04805712

INTERVENTIONS:
Drug: PF-04805712 — ascending single and multiple doses starting at 30 mg

SUMMARY:
To assess the safety and tolerability of escalating single and multiple doses of the compound in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of non-childbearing potential.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events, vital signs measurements, telemetry, 12 lead ECGs, blood and urine safety tests. | 12 weeks
Pharmacokinetics: PK parameters will be determined after single dose, fasted and (at one dose) fed, and at steady state (fasted or fed depending on single dose data). | 12 weeks

SECONDARY OUTCOMES:
Pharmacodynamics: Urinary LTE4 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1411001&StudyName=Single%20and%20multiple%20dose%20safety%2C%20tolerability%2C%20and%20pharmacokinetics%20study%20of%20PF-04805712%20in%20healthy%20volunteers